CLINICAL TRIAL: NCT04422223
Title: Copenhagen Liver Cohort Study: Disease Characteristics, Outcomes and Rehabilitation in Liver Cirrhosis - A Prospective Cohort Study
Brief Title: Prospective Cohort Study of Disease and Outcomes in Cirrhosis
Acronym: ProDoc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Nina Kimer, MD, PhD, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-19024348
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Liver Cirrhosis, Alcoholic; Progression; Liver Diseases; Decompensated Cirrhosis
Keywords: Prognosis; Prospective; Cirrhosis; Hepatology
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Disease Progression; Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma and buffy coat from whole blood, liver biopsies, stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients newly diagnosed with liver cirrhosis form the Gastro Unit, Amager Hvidovre Hospital, Denmark. All patients with clinically verified diagnosis, irrepsective of disease stage and etiology is included.

SUMMARY:
A population based incidence cohort will enroll patients newly diagnosed with cirrhosis to investigate disease characteristics and outcomes, explore mechanisms predicting early death and hospital admission, and assess new monitoring tools in treatment and prevention of cirrhosis.

DETAILED DESCRIPTION:
INTRODUCTION In Denmark the incidence of liver cirrhosis is increasing. From 1996 to 2005 the number of hospital admissions due to liver cirrhosis rose with 2,500 extra admissions per year. Patients who are readmitted to the hospital have a higher 90 days mortality than those who avoid readmission.

Liver cirrhosis in Denmark is caused by a wide use of alcohol and a population increasing in age and BMI.

The course of cirrhosis depends on etiology, age and nutritional status, as well as social factors such as personal network, employment and economy. Interventional studies on many of these mechanisms are still unexplored.

Cirrhosis is related to decreased quality of life and affects patients and relatives both emotional and socioeconomically.

The Gastro Unit, Amager Hvidovre Hospital has a catchment area of 550,000 citizens in South and West of Copenhagen. The Gastro Unit diagnoses app. 140 people with liver cirrhosis yearly.

Patient education and rehabilitation is implemented as standard health care after significant pulmonary or cardiac disease in all regions of Denmark.

HYPOTHESIS A systematic approach to investigation, treatment and rehabilitation in liver cirrhosis will improve the patient's ability to benefit from medical treatment and health care offers and increase patient involvement and autonomy in disease.

A systematic approach to investigation of liver disease will contribute to identify new risk factors for death, hospital admission and readmission, and decompensation in liver cirrhosis.

Better knowledge on sociodemographic features, use of health care resources and the patient's physical performance and frailty will improve new actions of personalized treatment, interventions focusing on patient needs and patient reported outcomes in cirrhosis.

Primary outcome The primary aim for this prospective cohort study is to improve characterization, treatment and rehabilitation under and after admission of patients with liver cirrhosis, with the purpose of improving survival and reducing risk of readmission.

Secondary outcomes

* To identify 'frail patients' and to improve their access to health care offers.
* To improve the utilization of health care resources by a systematic approach to patient characterization and treatment.
* To identify co-factors with importance for early death and readmission.
* To identify and explore new targets for treatment and symptom-relief in liver cirrhosis.

METHODS The cohort study will apply an observational prospective incidence cohort design in which patients will be followed from diagnosis to death or withdrawal from the cohort. Participants will be enrolled consecutively within six months of diagnosis.

TRIAL FLOW The standardized investigational program includes procedures recommended by National- and European guidelines for complications in liver cirrhosis, applied at the Gastro Unit, Medical Division, Amager Hvidovre Hospital.

The standard investigational program will be initiated within six months of inclusion. To avoid repetition of invasive diagnostic procedures (e.g. upper endoscopy, CT scan or ultrasound), we will accept retrospective inclusion of data, dating back to time of diagnosis (maximum six months).

Standard biochemistry will be performed at inclusion and at follow-up after 1,2,3 and 5 years.

Bio Impedance Assessment will be performed at inclusion and at follow up after 1,2,3 and 5 years.

Assessments of socio demography, loneliness and quality of life will be performed through the following questionnaires:

1. A specific questionnaire assessing socio demography, economic status and use of health care resources is designed for the trial.
2. Three item loneliness scale
3. Alcohol use by Audit C
4. Health related quality of life in cirrhosis by: Chronic Liver Disease Questionnaire (CLDQ).
5. Functional disability in work-, social- and family life by: Sheehan Disability Scale (SDS).

Information will be retrieved from the participant's medical record concerning:

* Dates and length of hospitalization.
* Reason for hospitalization.
* Diagnosis.
* Biochemistry.
* Results from endoscopic procedures.
* Results from ultrasound, CT scan, and if applied, MR scan.
* Results from Dexascan.

BIO BANK FOR FUTURE RESEARCH For this study a research bio bank for future research will be established. The bio bank will contain blood, liver tissue and stool.

The bio bank is registered separately by The Danish Data Protection Agency.

DATA A database in Redcap will be established for the study. Questionnaires will be answered electronically on an Ipad exporting data directly to Redcap. The Redcap database will use study ID numbers and initials for identification of participants. An identification list of all participants will be stored separately.

Investigators aim to publish all results derived from this trial. The investigators support open acces policy, and at the end of the trial, all data will be sought published in anonymous form.

ETHICS The study is approved by the Scientific Ethics Committees of the Capital Region of Denmark and The Danish Data Protection Agency before initiation.

A thorough characterization and consecutive inclusion will strengthen our knowledge on the incidence, prevalence and impact of liver disease in the population, and the use of health care resources allocated to liver disease.

The study will contribute to the finding of formerly unidentified risk factors with importance for survival and use of health care services; and thereby form the basis of implementation of changes in health practices, with both economic and medical gain. The study may also identify new areas for interventional research, with clinically relevant endpoints that can be translated into favorable changes in health care practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of cirrhosis supported by biochemistry and ultrasound or other imaging techniques.
* Cirrhosis of any etiology
* Informed written consent

Exclusion Criteria:

* People where the diagnosis of liver cirrhosis is questioned with reasonable doubt or the diagnosis of liver cirrhosis is disproved by histology or relevant imaging.
* Withdrawal of informed consent or no informed consent.
* Persons eligible for inclusion where the investigational program is delayed or not initiated within six months after the diagnosis of suspected cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a debut of liver cirrhosis, irrespective of time and circumstances of diagnosis, comorbidities and severity of disease will be offered inclusion in the cohort.
  A small percentage of patients will be diagnosed with cirrhosis at a very late stage of disease and have complications compromising their cognitive function. When complications are considered reversible, enrolment in the study will be sought when the patient has recovered. When complications are considered irreversible or there may be reasonable doubt of the patient's survival, patients will be considered eligible, but excluded to avoid unethical conduction of procedures.
  Participants may be diagnosed with terminal disease or end-stage liver disease. In such a case, to secure the integrity of the patient, no extra investigational procedures will be made and only data sampled in standard medical care will be used in the cohort database.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Improve risk of decompensation in cirrhosis | 5 years
  time to development of decompensation
Survival | 5 years
  Time from diagnosis to death or liver transplantation

SECONDARY OUTCOMES:
Risk prediction by Short Physical Performance Battery | 5 years
  Identify patients with low physical performance and assess their risk of decompensation and complications to liver cirrhosis
Characterization of patients | 5 years
  Describe characteristics of disease in the cohort
Social impact of cirrhosis | 5 years
  Assess the impact of social factors, use of health care ressources, including home nursing, with importance for early death and readmission
Life space Assessment | 5 years
  Evaluate mobility in cirrhosis by Life Space Assessment questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nina Kimer, Hvidovre, Please Enter the State Or Province, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We plan to share IPD in anonymuos form, in a data repository, possibly stored by the University of Copenhagen. Plans for the IPD derived from the biobank for future research will be made when protocols for these projects are completed.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5-10 years

REFERENCES:
- [Derived] Mynster Kronborg T, Webel H, O'Connell MB, Danielsen KV, Hobolth L, Moller S, Jensen RT, Bendtsen F, Hansen T, Rasmussen S, Juel HB, Kimer N. Markers of inflammation predict survival in newly diagnosed cirrhosis: a prospective registry study. Sci Rep. 2023 Nov 16;13(1):20039. doi: 10.1038/s41598-023-47384-2. PMID 37973887